CLINICAL TRIAL: NCT02240953
Title: Comparison of Different Anticoagulation Regiments in Patients With Prosthetic Heart Valve Non-ObstructiveThrombosis
Brief Title: Anticoagulation Regiments in Patients With Prosthetic Heart Valve Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MEHMET OZKAN, Principal Investigator, MD., Prof., Head of Cardiology, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOSUYOLU2
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Thrombosis
Keywords: Anticoagulation; Prosthetic Heart Valves; Acetylsalicylic acid; Warfarin; Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Warfarin (Active Comparator): In the first arm only warfarin is given with a target INR level of 2.5-4 to the patients with prosthetic heart valve thrombosis
  Interventions: Drug: Warfarin
- Warfarin + ASA 100 mg + PPI (Active Comparator): In the second arm 100 mg acetylsalicylic acid and a proton pump inhibitor are added to treatment in combination with warfarin for the patients with prosthetic heart valve thrombosis
  Interventions: Drug: Warfarin + ASA 100 mg + PPI
- Warfarin + ASA 300 mg + PPI (Active Comparator): In the third arm 300 mg acetylsalicylic acid and a proton pump inhibitor are added to treatment in combination with warfarin for the patients with prosthetic heart valve thrombosis
  Interventions: Drug: Warfarin + ASA 300 mg + PPI
- Observational Warfarin (Active Comparator): This arm is an observational group of patients who do not have prosthetic heart valve thrombosis. These patients also are followed under only warfarin therapy with INR level of 2.5-4.
  Interventions: Drug: Observational Warfarin

INTERVENTIONS:
Drug: Warfarin — Only warfarin is given with a target INR level of 2.5-4 to the patients with prosthetic heart valve thrombosis
  Arms: Warfarin
Drug: Warfarin + ASA 100 mg + PPI — 100 mg acetylsalicylic acid and a proton pump inhibitor are added to treatment in combination with warfarin for the patients with prosthetic heart valve thrombosis
  Arms: Warfarin + ASA 100 mg + PPI
Drug: Warfarin + ASA 300 mg + PPI — In the third arm 300 mg acetylsalicylic acid and a proton pump inhibitor are added to treatment in combination with warfarin for the patients with prosthetic heart valve thrombosis
  Arms: Warfarin + ASA 300 mg + PPI
Drug: Observational Warfarin — This is an observational group of patients who do not have prosthetic heart valve thrombosis. These patients also are followed under only warfarin therapy with INR level of 2.5-4.
  Arms: Observational Warfarin

SUMMARY:
Prosthetic valve thrombosis is a serious complication with high mortality and morbidity. However, the best anticoagulant treatment strategies for patients with prosthetic heart valve thrombosis have not been fully known. In this study the investigators wanted to identify the most effective and safe regimen among different anticoagulant regimens.

DETAILED DESCRIPTION:
Three different anticoagulant treatment regimens for patients with prosthetic heart valve non-obstructive thrombosis have been described. Patients are included in each group randomly. In the first arm only warfarin is given to the patients with a target INR level of 2.5-4. In the second arm 100 mg acetylsalicylic acid and a proton pump inhibitor are added to treatment in combination with warfarin. In the third arm 300 mg acetylsalicylic acid and a proton pump inhibitor are added to treatment in ombination with warfarin. Also there is an observational follow-up group of patients who do not have prosthetic heart valve thrombosis. These patients also are followed under only warfarin therapy with INR level of 2.5-4 . All patients are followed by serial transesophageal echocardiography performed every 6 months. Follow-up period is at least 6 months (range 6-60 months). Informed consent is taken from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prosthetic heart valve thrombosis

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Decreased thrombus size | 6 months
  Decreased thrombus size on control transesophageal echocardiography in the absence of fatal and non fatal major complications
Same thrombus size | 6 months
  Thrombus size remains as similar as the previous transesophageal echocardiographic examination findings in the absence of any fatal and non fatal major complications
Increased thrombus size | 6 months
  Increased thrombus size on control transesophageal echocardiography in the absence of fatal and non fatal major complications
Complications | 6 months
  Nonfatal major complication: Ischemic stroke, intracranial hemorrhage, embolism (coronary or peripheral), bleeding requiring transfusion
  Nonfatal minor complication: Bleeding without need for transfusion, TIA.

CONTACTS AND LOCATIONS:
Locations (1):
- Kosuyolu Kartal Heart Training and Research Hospital, Istanbul, Turkey (Türkiye)